CLINICAL TRIAL: NCT03117426
Title: A Randomised, Subject-masked Evaluation of Visual Function After Bilateral Implantation of Two Types of Presbyopia-correcting IOLs: the Symfony-study
Brief Title: A Randomised Evaluation of Visual Function After Bilateral Implantation of Two Types of Presbyopia-correcting IOLs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Abbott Medical Optics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NL56878.068.16
Record Dates: First submitted 2017-04-12; First posted 2017-04-18 (Actual); Last update posted 2018-05-02 (Actual); Status verified 2017-04

CONDITIONS: Cataract; Presbyopia
Keywords: Symfony Extended Range of Vision IOL; AT LISA tri 839MP IOL; Trifocal IOL; Extended depth of focus IOLs
MeSH Terms: conditions — Cataract; Presbyopia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SYMFONY IOL (Experimental): The unique design of this IOL merges two complementary enabling technologies: (1) its diffractive echelette design feature extends the range of vision, and (2) achromatic technology corrects chromatic aberration for enhanced contrast sensitivity. Theoretically, combining these two mechanism of action results in a continuous range of high-quality vision for far, intermediate, and near distances with the same low incidence of halos and glare associated with monofocal IOLs (see figure 2).
  Primary indication is implantation for the visual correction in adult patients in whom a cataractous lens has been removed, who desire useful vision over a continuous range of distances including far, intermediate, and near, resulting in spectacle independency. This device is intended to be placed in the capsular bag.
  Interventions: Device: SYMFONY IOL
- AT LISA tri 839MP IOL (Active Comparator): This trifocal IOL provides three useful focal distances, far, intermediate, and near, and therefore aims to provide functional visual restoration after cataract surgery.
  Primary indication is implantation for the visual correction in adult patients in whom a cataractous lens has been removed, who desire useful vision over a continuous range of distances including far, intermediate, and near, resulting in spectacle independency. This device is intended to be placed in the capsular bag.
  Interventions: Device: AT LISA tri 839MP IOL

INTERVENTIONS:
Device: SYMFONY IOL — IOL for presbyopic treatment in patients undergoing cataract surgery. EDOF IOL.
  Other Names: EDOF IOL
  Arms: SYMFONY IOL
Device: AT LISA tri 839MP IOL — IOL for presbyopic treatment in patients undergoing cataract surgery. Trifocal IOL
  Other Names: Trifocal IOL
  Arms: AT LISA tri 839MP IOL

SUMMARY:
Since the introduction of intraocular lenses (IOL) in the treatment of cataract, the postoperative accommodative loss of the human eye has been a trending topic. Numerous studies show a high rate of spectacle-independency after bilateral implantation of multifocal IOLs (MIOL). However, glare, halos, and reduced visual acuity under different light conditions are common complaints after MIOL implantation. Due to its unique design, the TECNIS® Symfony Extended Range of Vision ZXR00 IOL (Abbott Medical Optics, Santa Ana, USA, hereinafter referred to as Symfony IOL) is theoretically providing a continuous range of high-quality vision for far, intermediate, and near distances with the same low incidence of halos and glare associated with monofocal IOLs under different light conditions.

The goal of this study is to compare the AT LISA tri 839MP IOL (Carl Zeiss Meditec AG, Jena, Germany, hereinafter referred to as AT LISA IOL) versus the Symfony IOL in terms of postoperative achieved visual acuity at different distances, patient satisfaction (e.g. spectacle-independency, QoL), and postoperative complication profile (e.g. halo's and glare) under different light conditions. So far, there are no published studies comparing both IOLs. Therefore, we will perform this randomized control trial.

DETAILED DESCRIPTION:
Rationale: Since the introduction of intraocular lenses (IOL) in the treatment of cataract, the postoperative accommodative loss of the human eye has been a trending topic. Numerous studies show a high rate of spectacle-independency after bilateral implantation of multifocal IOLs (MIOL). However, glare, halos, and reduced visual acuity under different light conditions are common complaints after MIOL implantation. Due to its unique design, the TECNIS® Symfony Extended Range of Vision ZXR00 IOL (Abbott Medical Optics, Santa Ana, USA, hereinafter referred to as Symfony IOL) is theoretically providing a continuous range of high-quality vision for far, intermediate, and near distances with the same low incidence of halos and glare associated with monofocal IOLs under different light conditions.

The goal of this study is to compare the AT LISA tri 839MP IOL (Carl Zeiss Meditec AG, Jena, Germany, hereinafter referred to as AT LISA IOL) versus the Symfony IOL in terms of postoperative achieved visual acuity at different distances, patient satisfaction (e.g. spectacle-independency, QoL), and postoperative complication profile (e.g. halo's and glare) under different light conditions. So far, there are no published studies comparing both IOLs. Therefore, we will perform this randomized control trial.

Objective: The primary objective of this study is to compare the postoperative visual outcomes in a series of patients bilaterally implanted with the AT LISA IOL versus those bilaterally implanted with the Symfony IOL.

Study design: Single-centre randomised clinical trial. Study population: 30 patients (60 eyes) with bilateral cataract who require cataract surgery.

Intervention (if applicable): Cataract surgery with bilateral implantation of either a Symfony IOL or an AT LISA IOL.

Main study parameters/endpoints: The primary endpoint is the binocular uncorrected visual acuity at 66 cm distance under both photopic and mesopic conditions 13 weeks postoperatively. Secondary endpoints are: binocular (un)corrected visual acuity at far (4 meters) and near (40 cm) under both photopic and mesopic conditions, reading performance, patient satisfaction, and complication profile.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Both lens models used in this study are CE-marked and commercially available. The pre- and postoperatively examinations to be performed in this study are part of the regular medical treatment of patients with cataract who need cataract surgery. There is one more postoperative visit compared to standard cataract surgery. Potential risks, such as postoperative residual refractive error, halo's and glare, associated with multifocal IOL implantation are expected to be comparable or even lower after implantation of Symfony IOL. Spectacle-independency and high quality visual acuity postoperatively are the expected major benefits of implantation of the Symfony IOL.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 21 years of age
* Bilateral cataract
* Bilateral implantation of Tecnis Symfony IOL or AT LISA IOL (same lens model in both eyes)
* Expected postoperative astigmatism ≤ 1.00 D (combination with FLACS AK is tolerated up to 1.5 D preoperative astigmatism)
* IOL power calculation between +10.00 D and 32.00 D
* Expected postoperative best-corrected visual acuity of logMAR +0.3 or better
* Availability to undergo second eye surgery within 2 weeks of the first eye surgery
* Willing and able to comply with scheduled visits and other study procedures
* Signed informed consent.

Exclusion Criteria:

* Previous corneal surgery and/or reshaping
* Clinically significant corneal endothelial dystrophy (e.g., Fuchs' dystrophy)
* Irregular astigmatism
* Keratoconus
* History of corneal disease (e.g., herpes simplex, herpes zoster keratitis, etc.)
* Extensive age related macular degeneration (atrophic or exudative age-related macular degeneration or numerous soft drusen)
* Extensive visual field loss (e.g., glaucoma, history of cerebral vascular accidents, etc.)
* Extensive diabetic macular disease
* History of amblyopia and/or strabismus
* Pseudoexfoliation syndrome or other capsule or zonular abnormalities that could affect postoperative centration or tilt of the IOL
* Pupil abnormalities (non-reactive, tonic pupils, abnormally shaped pupils, or pupils that do not dilate at least 3.5 mm under mesopic/scotopic conditions)
* Cognitive, cerebral or concentration disorders (e.g. dementia, Parkinson, history of CVA, etc.)
* Suturing of incision required at time of surgery
* Complications during surgery of the first eye.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Binocular uncorrected intermediate (66cm) visual acuity under both photopic and mesopic conditions. | 3 months / 13 weeks
  The mean binocular uncorrected intermediate visual acuity at 66 cm under both photopic and mesopic conditions at 13 weeks (3 months) postoperatively

SECONDARY OUTCOMES:
Binocular visual acuity | 3 months / 13 weeks
  At 4 meter, 40 cm, including reading speed
Quality of Life | pre-op and 3 months/13 weeks
  QoL questionnaires
Contrast sensitivity | 3 months/13 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rudy Nuijts, MD PhD, Principal Investigator — University Eye Clinic Maastricht, Maastricht University Medical Centre
Locations (1):
- Maastricht University Medical Centre, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared